CLINICAL TRIAL: NCT07141511
Title: A Phase 1, Single-dose, Open-label, Randomized, Crossover Study in Healthy Adult Participants to Evaluate Relative Bioavailability and Food Effect of a Fixed-Dose Combination Tablet Containing Zanubrutinib and Sonrotoclax (BG-71332)
Brief Title: A Study to Investigate the Relative Bioavailability and Food Effect of a Fixed-Dose Combination Tablet Containing Zanubrutinib and Sonrotoclax (BG-71332) in Healthy Adults
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BeOne Medicines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: BG-71332-101
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BG-71332, Zanubrutinib + Sonrotoclax (Experimental): Participants will receive the following treatments in one of six sequences: one dose of BG-71332 with a high-fat meal, one dose of BG-71332 in a fasted state, and one dose of zanubrutinib and sonrotoclax administered together with a high-fat meal.
  Interventions: Drug: BG-71332; Drug: Zanubrutinib; Drug: Sonrotoclax

INTERVENTIONS:
Drug: BG-71332 — Administered orally
Drug: Zanubrutinib — Administered orally
  Other Names: BGB-3111
Drug: Sonrotoclax — Administered orally
  Other Names: BGB-11417

SUMMARY:
The purpose of this study is to evaluate the relative bioavailability of a fixed-dose combination tablet containing zanubrutinib and sonrotoclax (BG-71332) compared to a zanubrutinib capsule and sonrotoclax tablet administered simultaneously and the effect of food on how the body processes the fixed-dose combination tablet.

ELIGIBILITY:
Inclusion Criteria:

* In good health, determined by no clinically significant findings from medical history, 12-lead ECGs, vital sign measurements, and clinical laboratory evaluations as assessed by the investigator.
* An absolute B-cell count of >200 cells/μL.
* Female participants must be of non-childbearing potential (surgically sterile or postmenopausal).

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator or designee.
* Evidence of any infections (bacterial, viral, fungal, parasitic) within 4 weeks prior to the first dose of study drug, as determined by the investigator (or designee).

Note: Other protocol defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2025-09-24 (Actual); Primary Completion 2026-02-22 (Estimated); Study Completion 2026-02-22 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from time 0 extrapolated to infinity (AUC0-inf) for zanubrutinib | Predose and up to 72 hours post dose
Area under the plasma concentration-time curve from time 0 extrapolated to infinity (AUC0-inf) for sonrotoclax | Predose and up to 72 hours post dose
Area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration (AUC0-t) for zanubrutinib | Predose and up to 72 hours post dose
Area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration (AUC0-t) for sonrotoclax | Predose and up to 72 hours post dose
Maximum observed plasma concentration (Cmax) of zanubrutinib | Predose and up to 72 hours post dose
Maximum observed plasma concentration (Cmax) of sonrotoclax | Predose and up to 72 hours post dose

SECONDARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) | Up to 30 days after last dose, up to approximately 47 days
Number of participants with laboratory abnormalities | Up to 30 days after last dose, up to approximately 47 days
  Laboratory parameters include hematology, clinical chemistry, and urinalysis test results
Number of participants with clinically significant abnormal electrocardiogram (ECG) values | Up to 30 days after last dose, up to approximately 47 days
Number of participants with clinically significant vital signs measurements | Up to 30 days after last dose, up to approximately 47 days

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeOne Medicines
Locations (1):
- Linear Early Phase, Joondalup, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: Yes
BeOne shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeOne shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeOne review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beonemedicines.com/science/clinical-trials/